CLINICAL TRIAL: NCT06893627
Title: Body Project SMIL: Effectiveness of Virtually Delivered Body Project Groups to Prevent Eating Disorders Among Young Women With Psychiatric Illness
Brief Title: Body Project SMIL: Prevention of Eating Disorders Among Young Women With Psychiatric Illness With the Body Project
Acronym: BP_SMIL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Aalborg Psychiatric Hospital (Other)
Responsible Party: Principal Investigator, Loa Clausen, Ass. Prof. Psychologist, PhD, senior researcher, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1-10-72-71-24
Record Dates: First submitted 2025-03-11; First posted 2025-03-25 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Eating Disorders; Psychiatric Disorder; Body Dissatisfaction; Eating Disorder Symptom and Body Image Dissatisfaction
Keywords: Prevention of eating disorders; Dissonance-based prevention; psychiatric ilness
MeSH Terms: conditions — Feeding and Eating Disorders; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Body Project intervention (Experimental): Dissonance-based, online, peed-led intervetion, consisting of 4 x 1 hour with a week a part.
  Interventions: Behavioral: Body Project
- Expressive writing (Active Comparator): The expressive writing as the active control condition, will consist of written instructions sent to participants weekly over 4 weeks, asking them to write about their own thoughts or feelings in relation to their body for 40 min.
  Interventions: Behavioral: Expressive writing

INTERVENTIONS:
Behavioral: Body Project — Dissonance-based, online, peed-led eating disorder prevention intervention, consisting of 4 x 1 hour with a week a part.
  Arms: Body Project intervention
Behavioral: Expressive writing — Participants are encouraged to write about their body 40 min. per week
  Arms: Expressive writing

SUMMARY:
The Body Project SMIL tests the effectiveness of a virtual, peer-led intervention aimed at reducing body dissatisfaction and preventing eating disorders in young women with psychiatric illnesses.

Eating disorders like anorexia, bulimia, and binge eating disorder have severe physical and mental health consequences. Young women with psychiatric disorders face a fourfold higher risk, yet no widely implemented prevention programs exist in Denmark. Body Project SMIL addresses this gap by testing whether a structured online intervention can prevent eating disorders before they develop.

The study is open to women aged 15-25 with body dissatisfaction and a verified psychiatric diagnosis (e.g., mood disorders, anxiety, ADHD, or personality disorders). Those with a clinical eating disorder diagnosis are not eligible. Participants must be comfortable engaging in online group discussions.

Participants are randomly assigned to one of two groups:

Body Project Group - A peer-led, virtual program with four one-hour sessions focusing on challenging beauty ideals through structured exercises.

Expressive Writing Group - A self-guided exercise where participants write about body image for four weeks.

Assessments take place before and after the intervention, with follow-ups at six months, one year, and two years tracking body dissatisfaction, eating disorder symptoms, and well-being.

The Body Project is a proven intervention that reduces body dissatisfaction, thin-ideal internalization, and eating disorder symptoms, with some studies showing a 77% reduction in eating disorder risk. While tested in various settings, this study is the first to evaluate its impact on young women with psychiatric illnesses.

Participation benefits may include improved body image, reduced eating disorder risk, and enhanced self-esteem. The group format provides a supportive environment for sharing experiences and fostering healthier attitudes toward body image.

Ethical approval has been granted, ensuring compliance with GDPR regulations. Since this is a preventive program, it does not replace clinical treatment. Participants showing signs of an active eating disorder will be referred for appropriate care.

Recruitment occurs through psychiatric departments, educational institutions, and social media. A research website (www.bodyproject.dk) provides study details and a secure registration form. Parental consent is required for participants under 18, and all participants may withdraw at any time without consequences.

Conducted by Aarhus University Hospital Psychiatry in collaboration with international experts, this research may inform scalable prevention programs for young people at risk of eating disorders.

DETAILED DESCRIPTION:
Body Project SMIL:

Effectiveness of virtually delivered Body Project groups to prevent Eating Disorders among young Women with Psychiatric Illness (part of Body Project DK)

Background:

Eating disorders (ED) are characterized by extreme fear of weight gain, dietary restraint, binge eating, and compensatory behaviors such as self-induced vomiting, excessive exercise, and misuse of laxatives and diuretics with the main diagnostic categories being anorexia nervosa, bulimia nervosa, and binge eating disorder (DSM-5).

ED's are associated with functional impairment, reduced Quality-of-life, increased co-morbidity and mortality. Peak incidences for most ED are between the ages of 16 to 20 indicating that ED prevention initiatives should be implemented within this specific age group.

Health care costs for ED's, especially anorexia nervosa, are high, few receive diagnosis and treatment and among those who do less than 50% produce symptom remission. In addition, persons with binge eating disorders and bulimia nervosa usually go untreated for years or even decades. Thus, there is a need for effective evidence-based prevention programs to reduce future onset of ED in the general population, but especially in high-risk groups.

One of the most dominant risk factors, and primary drivers of eating disorders, is body dissatisfaction. Body dissatisfaction has been on the rise among adolescents the latter decades. Individuals with other primary disorders like psychiatric illness and chronic diseases have increased risk of eating disorders. The risks are 4-fold among those with psychiatric illness. For individuals with psychiatric illness the increased risk might be related to the elevated distress of interpersonal problems related to the primary disorder or shared genetic factors.

The Body Project:

The Body Project is a dissonance-based therapy to help participants understand how society and social media affect our perception of body and appearances. It is currently the most studied ED prevention program reducing ED symptoms and future onset of ED with up to 77% (relative risk) compared to control group.

The Body Project contain 4 1-hour group sessions led by facilitators and is mostly tested in females with body image concern. The program is developed at Stanford University, Oregon Research Institute, USA, by Professor Eric Stice. During and between sessions, participants are encouraged to engage in both verbally, written, and behavioral exercises critiquing the thin ideal in society. These activities result in a subsequently reduced endorsement of the thin-ideal due to the cognitive dissonance, motivating participators to alter their cognitions to restore consistency.

Body Project produce significantly greater reductions in thin-idealization, body dissatisfaction, dieting, negative affect, and ED symptoms compared to control groups among 15+ years females at post-test and at 2-3-year follow-up and risk of onset of obesity at 1-year follow-up, than control groups.

The Body Project is most effective in reducing the onset of new ED when facilitated, or co-facilitated, by peers.

A recent meta-analysis concluded that the peer-led in-person Body Project intervention reduced the future onset of eating disorders with 58% over a period of 4 years. The Body Project has not reduced future onset of ED when facilitated solely by clinicians. Health promotion interventions are perceived as more credible if delivered by individuals who are recognizable by participants. Previous studies have mostly been in-person, but recent studies point towards a similar efficacy when delivered online . A Swedish RCT documented that a virtually delivered peer-led Body Project intervention was superior to an expressive writing control group in preventing later ED onset, i.e. a relative risk reduction of 77% in the 2-year incidence of ED in the virtual Body Project group. To the best of investigators knowledge Body Project has not been tested in young females with psychiatric illness, despite the 4-fold increased risk of ED in this group.

Considering the significant physical and psychological impacts of EDs it is imperative that research focus on effective and implementable ED prevention. With 4 online sessions the Body Project is an easily accessible, scalable, and cost-effective approach to reduce the future incidence of ED and improve overall well-being among vulnerable adolescents in Denmark. The absence of ED prevention programs in general and across a specter of vulnerable young people in Denmark calls for action.

Objectives:

The present study aims to test the efficacy of the Body Project as a virtually delivered peer-led intervention including women with psychiatric illness and body dissatisfaction with outcomes outlined below..

Investigotors propose the following hypothesis across:

I. The Body Project intervention will be effective in reducing incidence of ED (primary outcome) over a 2-year period compared to controls.

II. The Body Project intervention will significantly reduce ED symptoms and body dissatisfaction and increase Quality-of-Life.

III. Associations between psychiatric symptoms, body dissatisfaction and eating disorder symptoms across the 2 years will be tested.

Additionally, we will update and include So-Me items into the Body Project manual introduction and test the effect of So-Me time on symptom level and outcome. Also, qualitatively studies on the group dynamics as a part of the efficacy counteracting loneliness and feeling different is expected.

Methods:

The present study applies a randomized control trial methodology.

Participants and procedure:

All participants will be self-referrals. Investigators will make information on the project available as leaflets, either in print or shared on social media (Instagram and TikTok). A specific research website (www.bodyproject.dk) will be established containing participant information and contacts. The specific wording in the recruitment "Do you want to beat your body dissatisfaction?" ("Overvind din kropsutilfredshed") will aid in the natural selection of women with high-risk. QR codes will be applied for leaflets and will link directly to the participant information sheet on the webpage. Investigators purposely do not make contact information available on the leaflet as investigators would like to nudge participants to the participant information on the webpage prior to contacting investigators. The webpage will contain the same participant information as included in this application, for participants and parents. In addition, a registration form for expression of interest will also be available.

Psychiatric Departments throughout Denmark can inform about the project and hand out the information leaflets. Information leaflets about the project will also be send to educational organizations (upper secondary schools, high schools, vocational educations,) in Region Midt and Region Nord for possible posting.

In- and exclusion criteria outlined below.

The participant information and information sent to parents are similar, except for added parental guidance on how best to support their adolescents.

Step-by-step recruitment procedure

1. Participants can scan the QR code and will be sent to the participant information on the website and here they can declare interest using a link to a secure REDCap survey where they can share contact information and give consent to receive at screening video call.
2. Subsequently participants will receive an invitation via secure mail including participant information and a personal link to a video call with a trained member of the research group. In addition, investigators will contact them by phone to remind them to attend the video call. For the video call participants are informed about the right to invite a parent or another support person, to attend with them. Participants are also advised to have read the participant information and receive the call in a private place. Eligibility for participation will be established following a project specific flowchart. In cases of eligibility, participants are informed in detail about the project, including purpose, procedures and expected outcomes.

   For participants between 15-17 years, both participants and parents will receive the written information and both participants and parents should be present for the video call. For participants between 15-17 years an informed parental consent is required. Parents are encouraged to discuss potential participation with their adolescents.
3. If the participant maintains interest in project during the video call, the participants (and parents in case participant is between 15-17 years) will receive written participant information and the consent form, signed by the healthcare professional who conducted the initial video call via secure mail, with a possibility of providing a digital consent (via REDCap). This ensures that the level of information is similar and that parents can guide their children in the decision. For those between 15-17 years, a digital consent will be obtained from parents and the adolescent. If the participant turns 18 years old during the project, she will be required to fill out a new consent.
4. After a written consent is received a copy of the consent is sent to the participant via secure mail.
5. After inclusion baseline data will be collected, including selected measurements (see below and attached) and the eating disorder diagnostic interview. The latter will be done using a video call. Participants presenting with a current ED will be excluded from the studies and advised to seek assistance with their general practitioner.
6. All remaining will be randomly assigned to one of the two interventions (Body Project or expressive writing) each lasting for 4 weeks.
7. Before and after the intervention each participant will be sent a secure link to the survey. This will be repeated at the end of intervention and ½, 1 and 2 years after inclusion. Filling in questionnaire is expected to take 15-20 minutes. At baseline and at 1- and 2-year follow-up a diagnostic interview will also be performed.

The intervention is minimally invasive as it solely includes group discussions and because the content is manual-based, no group member, nor facilitators are able to stray into potential unsafe directions. Previous Body Project trials have shown no adverse events. As mentioned, it is of minimally invasive character and all 4 online groups sessions will be executed in a psychologically safe environment as sessions are word-by-word scripted, peers thoroughly trained and supervised. The sessions do not include a focus on the psychiatric illness which is only seen as a vulnerability factor in terms of their risk of developing an eating disorder in the long term. If participants raise questions regarding these, they will be informed to contact their primary health care professionals, i.e. general practitioner, psychiatrist or psychologist. Instead, the focus of the groups is to discuss and challenge the body ideals they encounter in the daily lives of participants. If participants report a worsening of their psychiatric condition, they will be offered an individual talk after the group session to help them connect with their primary care providers. In addition, based on the procedure being by self-referral, investigators believe the adolescents elicit substantial personal resources and a commitment to actively work on body image issues. Having shown this initiative and resource, investigators believe they should have the right themselves to decide whether to participate or not, and that preventing them from this, will undermine participants individuality. Combining the active self-referral process with eligibility determined by an experienced health professional from the research team based on specific inclusion and exclusion criteria and informing parents of participants under 18 years, will target appropriate participants.

Power calculation:

The incidence of new onset of ED over a period of 2-years is determined via the Eating Disorder Diagnostic Interview (EDDI) at baseline and 1- and 2-year follow-up. Based on a previous study we expect significant differences between groups, with an incidence of ED in the control group of 8.8% and 2% in the intervention group. Investigators accept a significance level of 0.05 (α) and a power of 0.80 (β), leading to a sample size of 137 in each arm. To control for attrition, we aim to include 150 in each arm. Attrition rates have been reported as increasing with 12% at 2-years and 19% at 4 years-follow-up.

The Body Project Intervention:

Minor cultural or disease specific adaptations to the general Body Project manual will be made, in collaboration with Stice and including participants perspectives. Sessions are held via a secure online platform, uniquely applicable to invited participants. Decision of specific platform depends on advise for IT-security Region Midtjylland. Sessions are recorded as this will enable supervision and fidelity assurance to ensure compliance with the manual. Short individual follow-up contacts via phone and/or e-boks will be made if participants miss a session. Each group will consist of 6-8 group members as in previous studies. The groups are by led two peers. The peer is a trained young adult, i.e., a student within the area of health care (medicine, dietetics, psychology, nursing).

All facilitators will receive extensive and continuous training and supervision.. Fidelity assurance and continuous monitoring and evaluation of sessions will be performed in regular supervision. Previous fidelity testing has shown high inter-rater agreement for the original Body Project.

Active control intervention (Expressive writing):

The expressive writing (EW) as the active control condition, will consist of written instructions sent to participants weekly over 4 weeks, asking them to write about their own thoughts or feelings in relation to their body for 40 min. This version of EW was used as earlier trials has found them equally credible to the Body Project. The output is solely for the participants themselves and will not be read by others.

User involvement in project:

User involvement is planned from beginning of the project, as focus group meetings with 4-5 users elaborating on especially recruitment methods, retention, social media platforms, and cultural adjustment of the manual.

Measures:

Applying a methodology including selection of measurements from existing Body Project literature, will allow for comparison across studies thereby augmenting effect estimates. All questionnaires will be set up in REDCap and questionnaires still in English will be translated and back-translated according to guidelines.

Data analysis:

The primary outcome, number of ED cases, will be tested using Chi-square tests. Secondary outcomes of continuous variables will be investigated using t-test, and for categorical variables using Chi-square tests. Continuous data will be displayed as mean ± standard deviation (SD) and categorical data will be displayed as absolute numbers and percentages [n (%)]. A p-value <0.05 is considered statistically significant. Mixed effect models will be performed to investigate longitudinal changes in anthropometry and eating disorder symptoms from baseline to 6 months and baseline to 2 years. Multiple linear regression analysis adjusting for age will be performed to explore associations between baseline variables, post measurement, 6, 12 months and, 1- and 2-years post-intervention on ED symptomology.

Regression analysis will be used to explore potential predictors of ED symptom reduction e.g. zBMI, so-me use, degree of psychiatric disorder load.

Research group, organization and collaborations:

The SMIL Project will be conducted from Department of Child and Adolescent Psychiatry, Aarhus University Hospital Psychiatry but is developed in collaboration with Steno Diabetes Center Aarhus. Both departments are experienced in conducting RCT's and have high level international educational environment for the PhD candidates.

Research group will consist of PI: PhD. Ass. Prof. Loa Clausen, Department of Child and Adolescent Psychiatry, Research Unit, Aarhus University Hospital Psychiatry with 25 years in the eating disorder field and Co-PI and coordinator: Phd. Stud. Cl. dietician, Master in pedagogical psychology, Caroline Bruun Abild, Steno Diabetes Center Aarhus, Aarhus University Hospital with several years of clinical and research experience with (disturbed) eating behaviors. The project is planned to include one PhD student and one post-doctoral position as Co-PI and coordinator (Caroline Bruun Abild).

An advisory board meeting 1-2 times a year includes a broad range of researchers with expertise in conducting RCT's and epidemiological studies, as well as research and clinical experience within the fields of ED, obesity, diabetes. Also, stakeholders representing patient organizations and users of BP will be invited.

Identified representatives includes:

Professor, MD, Eric Stice, Stanford University, author of The Body Project and +100 papers on ED prevention, PhD. Psychologist, Line Wisting, PI on multi-site Body Project Study, Oslo University Hospital, Professor, MD, Jens Meldgaard Bruun, Aarhus University, professor of clinical nutrition with a wide knowledge with both treatment and prevention of obesity and extensive research experience in conducting large randomized controlled trials, Professor Annelli Sandbæk, Aarhus University, professor in general medicine with a special focus on health care of adolescents across sectors.

Gry Kjærsdam Telléus, PhD psychologist, Department of Psychiatry Research, Aalborg University.

Perspectives:

This study will build on a large scale of international Body Project studies and contribute with knowledge of the effect on a specific high-risk group that have not been tested before. As no prevention programs exist in Denmark the project has, if results are satisfying, potential to be up-scaled to a national set-up. With low cost and the promising results from prior studies this could have tremendous national effect, both on the QoL in individuals with increased body dissatisfaction but also on national health care cost related to individuals with eating disorders. As no one has tested the Body Project in young women with psychiatric illness this study fill a gap in the internationals research on the prevention of eating disorders.

Ethical considerations:

The study conforms to the Declaration of Helsinki, and the protocol is registered at the Danish data protection agency at Region Midtjylland. Since some of the participants are under 18 years old, all information related to the study has been tailored for this age group and has included representatives from this demographic in the testing process. Before including participants, information of purpose, and potential risks or benefits of the study are given to all participants at the initial interview and afterward in written form to both participants and participants parents (if participants are between 15 and 17 years) via secure mail. All participants are provided a window of opportunity (minimum 24 hours) to consider participation. If they choose to proceed a written informed consent is obtained from all participants via RedCap as described in the section "Participants and procedure". Participants between 15 and 17 years will need parent consent besides participants own.

All data will be stored in a Redcap database at Aarhus University securing the General Data Protection Regulation.

Risk of adverse events:

With reference to the extensive previous Body Project literature, both including the virtual delivery mode and peer led interventions, investigators consider Body Project to be safe and applicable for this project. Investigators do not expect any adverse events due to participant in the Body project DK as this has not previously been reported in similar settings, we will however continuously monitor participants on several parameters, and register any adverse events, which will be discussed, and appropriate action will be taken. As this is an ED prevention program targeting individuals with body dissatisfaction, participants with a current ED diagnosis will be excluded from the study and advised on treatment options.

ELIGIBILITY:
Inclusion Criteria:

* self-reported body dissatisfaction and a medically verified psychiatric diagnosis (e.g., mood disorders, anxiety disorders, ADHD, and personality disorders)

Exclusion Criteria:

* ED symptoms equivalent to clinically significant ED corresponding to a diagnostic level according to DSM-5 criteria as evaluated via the Eating Disorder Diagnostic Interview.
* Acute psychiatric instability or psychosis or suicide attempt within the last 12 months, or inability to cognitively understand the project or work in the online group setting either due to illness or severe substance abuse.
* Not speaking and understanding Danish.

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Eating Disorders | Baseline, 1 year and 2 years
  Prevalence of clinical eating disorders. The semi-structured Eating Disorder Diagnostic Interview (EDDI) assesses ED symptoms including binge eating and purging corresponding to DSM-5 ED diagnoses, and will be used to determine anorexia nervosa, bulimia nervosa, binge eating disorder, and purging disorder.
  EDDI is a structured diagnostic interview assessing DSM-5 eating disorder criteria, yielding presence/absence of diagnoses and symptom frequency/severity.

SECONDARY OUTCOMES:
Eating Disorder symptoms | Baseline, 1 month, 1/2 year, 1 year, 2 years
  Prevalence of binge eating disorder symptoms according to Eating Disorder Examination Questionnaire (EDE-Q). EDE-Q is a self-report version of the Eating Disorder Examination, item 13-15, including frequency of behavior.
Eating Disorder symptoms | Baseline, 1 month, 1/2 year, 1 year, 2 years
  Prevalence of eating disorder symptoms and disordered eating behaviors according to Dutch Restraint Eating (DRES)Scale containing 10 items.
  Min. 11 - max. 50 ( lower scores indicate greater pathology)
Thin-idealization | Baseline, 1 month, 1/2 year, 1 year, 2 years
  The 8-item Ideal-Body Stereotype Scale-Revised assesses pursuit of the thin ideal (IBSSR).
  Min. 8- max. 40 (lower scores indicate greater body dissatisfaction)
Body Dissatisfaction and overevaulation of body and shape | Baseline, 1 month, 1/2 year, 1 year, 2 years
  The 10-item Body Dissatisfaction Scale assesses dissatisfaction with various body part.
  Min. 11 - max. 50 ( lower scores indicate greater dissatisfaction)
Overevaluation og appearence, weight and shape | Baseline, 1 month, 1/2 year, 1 year, 2 years
  Overevaluation of appearance, weight and shape will be measured by three items inspired by the Eating Disorder Examination Questionnaire (EDE-Q) item number 22 + 23, min. 0-max. 12 (greater scores indicate greater pathology)
Substance use | Baseline, 1 month, 1/2 year, 1 year, 2 years
  Substance use are measured by three questions:
  How many times per week do you drink alcoholic beverages? How many times per week do you smoke (cigarettes, e-cigarettes, puff bars) or use nicotine products? How many times per week do you use recreational drugs? (e.g., cannabis, cocaine, psychedelic substances, etc.)
Loneliness | Baseline, 1 month, 1/2 year, 1 year, 2 years
  Loneliness will be assessed through Brief Symptom Inventory (BSI) item 5. rated on a 5-point scale (0-4), with higher scores indicating greater loneliness
Anxiety symptoms | Baseline, 1 month, 1/2 year, 1 year, 2 years
  Anxiety symptoms (symptoms of generalized anxiety disorder) as anxiety experienced within the past 14 days was measured using The Generalized Anxiety Disorder 2-item (GAD-2) scale Min. 0-max. 6 (greater scores indicate pathology)
Functional Impairment | Baseline, 1 month, 1/2 year, 1 year, 2 years
  Functional Impairment will be examined using the Clinical Impairment Assessment (CIA), which examines the psycho-social impairment due to eating disorder symptoms. The CIA is a 16-item, self-report questionnaire rated on a 4-point Likert-like scale, ranging from 0 ("Not at all") to 3 ("A Lot").
  Min. 0- max. 48 (greater scores indicate greater pathology)
Depression symptoms | Baseline, 1 month, 1/2 year, 1 year, 2 years
  Depression experienced within the past 14 days will be measured using the Patient Health Questionnaire (PHQ-2) scale 2 items min. 0-max 6 (greater scores indicate greater pahtology)
Positive and Negative affect | Baseline, 1 month, 1/2 year, 1 year, 2 years
  Positive and Negative affect, will be assessed using The Positive and Negative Affect Schedule Short Form (PANAS SF) 20 items, min 20- max 100 (greater scores indicate greater pathology)
Stress | Baseline, 1 month, 1/2 year, 1 year, 2 years
  Stress will be assessed using the single-item: "How often do you feel stressed?"
Psychological distress | Baseline, 1 month, 1/2 year, 1 year, 2 years
  Psychological distress, will be assessed using Brief Symptoms Inventory 18 (BSI-18), 18 items, min. 18- max. 90 (greater scores indicate greater pathology)
Physical activity | Baseline, 1 month, 1/2 year, 1 year, 2 years
  Physical activity wil be measured by one single question "How many hours per week are you physicallt active?"
Sleep problems | Baseline, 1 month, 1/2 year, 1 year, 2 years
  Sleep problems will be measured by a single question: "Within the past 6 months, how often have you had sleep problems?"
Social media use | Baseline, 1 month, 1/2 year, 1 year, 2 years
  Social media use will be assessed with multiple items to create two distinct social media use measures, evaluating what influence the respective platforms had on their body perception:
  How many hours per week do you spend on social media? How many hours do you spend on each social media (TikTok, Instagram, Facebook, Snapchat, Pinterest, other) How do the social media affect body perception (no impact, positive impact, negative impact, both positive and negative impact)
Health Care Utilization | Baseline, 1 year and 2 years
  Health Care Utilization, during the past 1 months will be assessed using two items: 1) the number of times participants saw a general practitioner, a private psychologist/psychiatrist or a health care professional in psychiatry, or another person because of physical or psychological illness, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Loa Clausen, PhD, Principal Investigator — Aarhus University Hospital Psychiatry; Caroline B Abild, Cl. dietician, Study Director — Aarhus University Hospital Psychiatry
Locations (1):
- Aarhus University Hospital Psychiatry, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Strien, T., et al., The predictive validity of the Dutch restrained eating scale. International journal of eating disorders, 1986. 5(4): p. 747-755.
- [Background] Wilfley DE, Schwartz MB, Spurrell EB, Fairburn CG. Assessing the specific psychopathology of binge eating disorder patients: interview or self-report? Behav Res Ther. 1997 Dec;35(12):1151-9. PMID 9465449
- [Background] Byrd-Bredbenner C, Eck K, Quick V. GAD-7, GAD-2, and GAD-mini: Psychometric properties and norms of university students in the United States. Gen Hosp Psychiatry. 2021 Mar-Apr;69:61-66. doi: 10.1016/j.genhosppsych.2021.01.002. Epub 2021 Jan 9. PMID 33571925
- [Background] Reas DL, Ro O, Kapstad H, Lask B. Psychometric properties of the clinical impairment assessment: norms for young adult women. Int J Eat Disord. 2010 Jan;43(1):72-6. doi: 10.1002/eat.20653. PMID 19260038
- [Background] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691
- [Background] Hovmand OR, Reinholt N, Christensen AB, Eskildsen A, Bach B, Arendt M, Poulsen S, Hvenegaard M, Arnfred SM. Affectivity in danish patients with emotional disorders: assessing the validity of the Positive and Negative Affect Schedule (PANAS). BMC Psychiatry. 2023 Dec 13;23(1):943. doi: 10.1186/s12888-023-05450-z. PMID 38093282
- [Background] Andersen S, Davidsen M, Nielsen L, Tolstrup JS. Mental health groups in high school students and later school dropout: a latent class and register-based follow-up analysis of the Danish National Youth Study. BMC Psychol. 2021 Aug 18;9(1):122. doi: 10.1186/s40359-021-00621-7. PMID 34407891
- [Background] Franke GH, Jaeger S, Glaesmer H, Barkmann C, Petrowski K, Braehler E. Psychometric analysis of the brief symptom inventory 18 (BSI-18) in a representative German sample. BMC Med Res Methodol. 2017 Jan 26;17(1):14. doi: 10.1186/s12874-016-0283-3. PMID 28125960
- [Background] Weissman MM, Bothwell S. Assessment of social adjustment by patient self-report. Arch Gen Psychiatry. 1976 Sep;33(9):1111-5. doi: 10.1001/archpsyc.1976.01770090101010. PMID 962494
- [Background] Stice E, Shaw H, Becker CB, Rohde P. Dissonance-based Interventions for the prevention of eating disorders: using persuasion principles to promote health. Prev Sci. 2008 Jun;9(2):114-28. doi: 10.1007/s11121-008-0093-x. Epub 2008 May 28. PMID 18506621
- [Background] Wisting L, Haugvik S, Wennersberg AL, Hage TW, Stice E, Olmsted MP, Ghaderi A, Brunborg C, Skrivarhaug T, Dahl-Jorgensen K, Ro O. Feasibility of a virtually delivered eating disorder prevention program for young females with type 1 diabetes. Int J Eat Disord. 2021 Sep;54(9):1696-1706. doi: 10.1002/eat.23578. Epub 2021 Jul 10. PMID 34245038
- [Background] Stice E, Rohde P, Shaw H, Gau JM. Clinician-led, peer-led, and internet-delivered dissonance-based eating disorder prevention programs: Effectiveness of these delivery modalities through 4-year follow-up. J Consult Clin Psychol. 2020 May;88(5):481-494. doi: 10.1037/ccp0000493. Epub 2020 Feb 24. PMID 32091226
- [Background] Festinger, L., A theory of cognitive dissonance. A theory of cognitive dissonance. 1957: Stanford University Press. xi, 291-xi, 291.
- [Background] Stice, E., P. Rohde, and H. Shaw, The Body Project: A Dissonance-Based Eating Disorder Prevention Intervention. 2012: Oxford University Press.
- [Background] Stice E, Onipede ZA, Marti CN. A meta-analytic review of trials that tested whether eating disorder prevention programs prevent eating disorder onset. Clin Psychol Rev. 2021 Jul;87:102046. doi: 10.1016/j.cpr.2021.102046. Epub 2021 May 21. PMID 34048952
- [Background] Ghaderi A, Stice E, Andersson G, Eno Persson J, Allzen E. A randomized controlled trial of the effectiveness of virtually delivered Body Project (vBP) groups to prevent eating disorders. J Consult Clin Psychol. 2020 Jul;88(7):643-656. doi: 10.1037/ccp0000506. PMID 32551736
- [Background] Barakat S, McLean SA, Bryant E, Le A, Marks P; National Eating Disorder Research Consortium; Touyz S, Maguire S. Risk factors for eating disorders: findings from a rapid review. J Eat Disord. 2023 Jan 17;11(1):8. doi: 10.1186/s40337-022-00717-4. PMID 36650572
- [Background] Momen NC, Plana-Ripoll O, Yilmaz Z, Thornton LM, McGrath JJ, Bulik CM, Petersen LV. Comorbidity between eating disorders and psychiatric disorders. Int J Eat Disord. 2022 Apr;55(4):505-517. doi: 10.1002/eat.23687. Epub 2022 Jan 27. PMID 35084057
- [Background] Conviser JH, Fisher SD, McColley SA. Are children with chronic illnesses requiring dietary therapy at risk for disordered eating or eating disorders? A systematic review. Int J Eat Disord. 2018 Mar;51(3):187-213. doi: 10.1002/eat.22831. Epub 2018 Feb 22. PMID 29469935
- [Background] Ottesen MA, A.A., Dahl KM, Lausten M, Boe Rayce S, Bille Tagmose B, BØRN OG UNGE I DANMARK - VELFÆRD OG TRIVSEL 2022. 2022.
- [Background] Austin A, Flynn M, Richards K, Hodsoll J, Duarte TA, Robinson P, Kelly J, Schmidt U. Duration of untreated eating disorder and relationship to outcomes: A systematic review of the literature. Eur Eat Disord Rev. 2021 May;29(3):329-345. doi: 10.1002/erv.2745. Epub 2020 Jun 23. PMID 32578311
- [Background] Helverskov JL, Clausen L, Mors O, Frydenberg M, Thomsen PH, Rokkedal K. Trans-diagnostic outcome of eating disorders: A 30-month follow-up study of 629 patients. Eur Eat Disord Rev. 2010 Nov-Dec;18(6):453-63. doi: 10.1002/erv.1025. PMID 20593480
- [Background] Hay P. A systematic review of evidence for psychological treatments in eating disorders: 2005-2012. Int J Eat Disord. 2013 Jul;46(5):462-9. doi: 10.1002/eat.22103. PMID 23658093
- [Background] Wonderlich SA, Peterson CB, Crosby RD, Smith TL, Klein MH, Mitchell JE, Crow SJ. A randomized controlled comparison of integrative cognitive-affective therapy (ICAT) and enhanced cognitive-behavioral therapy (CBT-E) for bulimia nervosa. Psychol Med. 2014 Feb;44(3):543-53. doi: 10.1017/S0033291713001098. Epub 2013 May 23. PMID 23701891
- [Background] Solmi M, Radua J, Olivola M, Croce E, Soardo L, Salazar de Pablo G, Il Shin J, Kirkbride JB, Jones P, Kim JH, Kim JY, Carvalho AF, Seeman MV, Correll CU, Fusar-Poli P. Age at onset of mental disorders worldwide: large-scale meta-analysis of 192 epidemiological studies. Mol Psychiatry. 2022 Jan;27(1):281-295. doi: 10.1038/s41380-021-01161-7. Epub 2021 Jun 2. PMID 34079068
- [Background] Klump KL, Bulik CM, Kaye WH, Treasure J, Tyson E. Academy for eating disorders position paper: eating disorders are serious mental illnesses. Int J Eat Disord. 2009 Mar;42(2):97-103. doi: 10.1002/eat.20589. No abstract available. PMID 18951455
- [Background] Stice E, Marti CN, Rohde P. Prevalence, incidence, impairment, and course of the proposed DSM-5 eating disorder diagnoses in an 8-year prospective community study of young women. J Abnorm Psychol. 2013 May;122(2):445-57. doi: 10.1037/a0030679. Epub 2012 Nov 12. PMID 23148784
- [Background] Koreshe E, Paxton S, Miskovic-Wheatley J, Bryant E, Le A, Maloney D; National Eating Disorder Research Consortium; Touyz S, Maguire S. Prevention and early intervention in eating disorders: findings from a rapid review. J Eat Disord. 2023 Mar 10;11(1):38. doi: 10.1186/s40337-023-00758-3. PMID 36899428
- [Background] Arcelus J, Mitchell AJ, Wales J, Nielsen S. Mortality rates in patients with anorexia nervosa and other eating disorders. A meta-analysis of 36 studies. Arch Gen Psychiatry. 2011 Jul;68(7):724-31. doi: 10.1001/archgenpsychiatry.2011.74. PMID 21727255
- See also: Body Project website including participant information — https://www.bodyproject.dk/